CLINICAL TRIAL: NCT01430533
Title: A Randomized, Double-blind, Vehicle Controlled Phase 1 Dermal Safety Study to Evaluate the Sensitizing Potential of Topically Applied Azelaic Acid Pre-foam Formulation in Healthy Subjects Using a Human Repeated Insult Patch Test Design
Brief Title: Human Repeated Insult Patch Test (HRIPT) of Azelaic Acid Pre Foam Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15854; 1401842 (Other: Company Internal)
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2014-02

CONDITIONS: Healthy
Keywords: dermal sensitization potential
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Verum (Experimental): Topical application of verum (azelaic acid pre foam formulation) on the skin
  Interventions: Drug: azelaic acid pre foam formulation
- Vehicle (Placebo Comparator): Topical application of vehicle formulation (same as verum but without active drug substance) on the skin
  Interventions: Drug: Vehicle pre foam formulation
- Negative control (Placebo Comparator): Topical application of distilled water (negative control) on the skin
  Interventions: Drug: Water

INTERVENTIONS:
Drug: azelaic acid pre foam formulation
  Arms: Verum
Drug: Vehicle pre foam formulation
  Arms: Vehicle
Drug: Water
  Arms: Negative control

SUMMARY:
The purpose of this study is to determine the dermal sensitization potential of azelaic acid pre-foam formulation.

DETAILED DESCRIPTION:
In an induction phase a three times weekly exposure over three weeks will be performed, followed by a resting phase. In a following challenge phase single exposure will be performed again and potential skin reactions observed. If skin reactions occur an optional re-challenge phase may be performed.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* male or female subjects
* aged 18 - 65 years
* ability to understand and fulfill the study requirements

Exclusion Criteria:

* affected skin in designated test area
* pregnancy or lactation
* not willing to comply with study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
skin sensitization reaction | day 3 to 6 of challenge phase week (week 6 or later, at least 2 weeks after the 3 week induction phase)
  skin reactions will be assessed, using a standardized scoring scale

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Robert I. Cooper, MD, Fargo, North Dakota, United States